CLINICAL TRIAL: NCT03954015
Title: Contrast Enhanced Ultrasound (CEUS) With US Microvessel Imaging, Contrast Enhanced Dual Energy Mammography (CEDM) and Contrast Enhanced Breast MR (CEMR): Comparison of Three Methods for Early Detection of Breast Cancer
Brief Title: Comparison of Three Methods for Early Detection of Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Katrina N. Glazebrook, M.B., Ch.B., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-003544
Record Dates: First submitted 2019-03-05; First posted 2019-05-17 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Proliferative Breast Disease
MeSH Terms: interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- patients over age 30 with suspicious BIRADS 4/5 Lesions (Other): Patients who are scheduled to undergo biopsy will be recruited to undergo imaging evaluation with CEDM, CEMR and CEUS.
  Interventions: Diagnostic Test: Contrast Enhanced imaging; Drug: Lumason

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced imaging — Contrast Enhanced Ultrasound (CEUS) with US Microvessel Imaging, Contrast Enhanced Dual Energy Mammography (CEDM) and Contrast Enhanced Breast MR (CEMR): Comparison of Three Methods for Early Detection of Breast Cancer.
  Other Names: Lumason
Drug: Lumason — FDA approved and used routinely for ultrasound exams of the heart and liver as well as the urinary tract in children. It contains microbubbles that are small enough to pass through the blood stream.

SUMMARY:
Subjects with suspicious breast lesion (BIRADS category 4/5) who are scheduled to undergo biopsy will be recruited to undergo imaging evaluation with Contrast Enhanced Dual Energy Mammography (CEDM), Contrast Enhanced Breast MR (CEMR) and Contrast Enhanced Ultrasound (CEUS).

DETAILED DESCRIPTION:
The co-primary endpoints are to estimate the sensitivity and specificity of CEUS relative to pathology determined diagnosis.

1. Positive predictive value of CEDM in detecting lesions seen on MR
2. Estimate the negative predictive value (TN/(TN+FN)) of CEUS as an adjunct.
3. Compare the frequency of recommendation of biopsy of MG±US vs MG±US plus CEUS as an adjunct based on BIRADS scores.
4. Comparison of background enhancement seen on CEUS with that seen on CEDM and CEMR.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Patients, greater than 30 years of age
* In good general health as evidenced by medical history
* BIRADS 4 or 5 suspicious breast lesions who are scheduled for breast biopsy.

Exclusion Criteria:

* Patients who are less than 30 years of age
* Have known or suspected cardiac shunts
* Have history of hypersensitive allergic reactions to any imaging contrast agents
* Pregnant (a urine pregnancy test will be given at no cost to the patient)
* Are nursing babies
* Poor renal function
* Are unwilling or unable (such as having a pacemaker) to undergo a CEMR

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females greater than 30 years of age
Enrollment: 3 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
CEUS true positive diagnosis | 1 year
  The number of CEUS true positive diagnosis defined as suspicious enhancement/ mass corresponding to area of malignant pathology at the time of biopsy based on lesion biopsy recommendation from diagnostic mammogram.
CEUS false positive diagnosis | 1 year
  The number of CEUS false positive diagnosis defined as suspicious enhancement corresponding to area of benign pathology at the time of biopsy based on lesion biopsy recommendation from diagnostic mammogram
CEUS true negative diagnosis | 1 year
  The number of CEUS true negative diagnosis defined as no enhancement corresponding to area of malignant pathology at the time of biopsy based on lesion biopsy recommendation from diagnostic mammogram.
CEUS false negative diagnosis | 1 year
  The number of CEUS false negative diagnosis defined as no enhancement corresponding to area of benign pathology at the time of biopsy based on lesion biopsy recommendation from diagnostic mammogram.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina N. Glazebrook, M.B., Ch.B., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials